CLINICAL TRIAL: NCT06801561
Title: EVALUATION of PREVENTIVE EFFECT of SEALANTS and LASER THERAPY on DENTAL CARIES and POSTERUPTIVE BREAKDOWN on MOLARS AFFECTED with MOLAR INCISOR HYPOMINERALISATION (RANDOMIZED CLINICAL TRIAL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Baraka, Lecturer, Pediatric dentistry department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AlexU-MB-MIH
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralisation; laser; sealant
MeSH Terms: conditions — Molar Hypomineralization | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): This group will be subjected to laser therapy. Er,Cr:YSGG will be used (Waterlase®, Biolase, USA) of a wavelength of 2780 nm at a power of 0.75 W using a frequency of 20 Hz and pulse duration of 140 µs. Irradiation will be performed on the entire occlusal and at the hypomineralized areas. The laser tip will pass in a uniform scanning motion steadily for 20 sec with relative isolation with 11% air and no water-cooling system. During the laser treatment, all safety measures will be followed.
  Interventions: Procedure: Laser therapy
- Control group (Active Comparator): This group will receive glass ionomer sealant. Conditioning of the surface will be done using polyacrylic acid (10%) conditioner for 20 seconds, then rinsed and dried. Fuji triage will be applied after activating and mixing the capsule. Light cure for 20 seconds. Occlusion will be checked using articulating paper and necessary adjustments will be done using finishing burs.
  Interventions: Procedure: Glass ionomer sealant

INTERVENTIONS:
Procedure: Laser therapy — This group will be subjected to laser therapy. Er,Cr:YSGG will be used (Waterlase®, Biolase, USA) of a wavelength of 2780 nm at a power of 0.75 W using a frequency of 20 Hz and pulse duration of 140 µs. (33) Irradiation will be performed on the entire occlusal and at the hypomineralized areas. (34) The laser tip will pass in a uniform scanning motion steadily for 20 sec with relative isolation with 11% air and no water-cooling system. During the laser treatment, all safety measures will be followed.
  Arms: Test group
Procedure: Glass ionomer sealant — This group will receive glass ionomer sealant. Conditioning of the surface will be done using polyacrylic acid (10%) conditioner for 20 seconds, then rinsed and dried. Fuji triage will be applied after activating and mixing the capsule. Light cure for 20 seconds. Occlusion will be checked using articulating paper and necessary adjustments will be done using finishing burs.
  Arms: Control group

SUMMARY:
Background: Molar Incisor Hypomineralisation (MIH) is a qualitative defect of enamel that shows asymmetrical involvement of one to four permanent first molars (PFM) with or without incisor teeth involvement. MIH molars are prone to post-eruptive breakdown (PEB) and to the development of atypical caries lesions.

Aim of the study: To evaluate and compare the preventive effect of glass ionomer sealant and laser therapy (LT) against dental caries and PEB on molars affected by molar incisor hypomineralisation (MIH) Materials and Method: This study is a two-arm, parallel group, randomized clinical trial. A sample of children (n=134) with an age range of 6-9 years old, having a first permanent molar erupted with MIH without PEB or carious lesion, will be selected from the outpatient clinic of Pediatric Dentistry and Public Health Department, Faculty of Dentistry, Alexandria University after securing necessary consents. All selected 134 first permanent molars will be randomly and equally allocated into two groups. Group 1(n=67): LT and Group 2 (n=67): Glass ionomer sealant (Fuji triage). Dental caries, PEB, retention of sealant and child-self-reported discomfort will be clinically evaluated after 6, 12 and 18months. Associations between dental caries and PEB with independent variables will be evaluated using logistic regression analysis (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* 6-9 years old children (29)
* One tooth with MIH with no PEB according to evaluation criteria proposed by Ghanim (2017) (APPENDIX I) (30) and ICDAS scores 0, 1 and 2 (APPENDIX II) (31)
* Good overall health (ASA I) (APPENDIX III) (32)

Exclusion Criteria:

* First permanent molars with active carious lesions with ICDAS scores 5 and 6 (Appendix II) or defective restorations (31)
* Sufficient dentin loss that requires restorative therapy
* Any clinical signs of failure (abscess, fistula)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Post-eruptive breakdown / dental caries | 21 months
  Initially, two examiners (MB and GW) will be pre-trained and calibrated to perform the MIH diagnosis based on the criteria described by Ghanim (2017). and ICDAS

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt